CLINICAL TRIAL: NCT03837054
Title: Does Chemotherapy Train the Mutation of the Pig-A Gene?
Brief Title: Does Chemotherapy Train the Mutation of the Pig-A Gene? (PIGA)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-63
Record Dates: First submitted 2019-01-16; First posted 2019-02-11 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Breast Cancer Female
MeSH Terms: interventions — Culture Techniques

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast cancer patients with external polychemotherapy (Other)
  Interventions: Biological: Blood collection and Micronuclei assay on binucleate lymphocytes in culture

INTERVENTIONS:
Biological: Blood collection and Micronuclei assay on binucleate lymphocytes in culture — The activity of the oncology Department of the North Hospital ensures the quick and easy recruitment of 30 patients over the 10-month inclusion period. The collection of samples will be done in a forward-looking manner during chemotherapy and at different times. The patients will have 4 blood samples of 10 mL carried out during their chemotherapy with a sampling at T0 (before the initiation of chemotherapy), then to T1 (after the first 3 cures), to T2 (after the 6th cure) and to T3 is 5 weeks after the end of the chemo And before the onset of radiation therapy. The samples will be carried out within the Medical Oncology Department of the hospital Nord of Marseille.
  We will also perform micronuclei testing on Binucleate lymphocytes in culture. The lymphocyte Micronuclei test reveals structure and number chromosomal damage and allows to reveal clastogenic or eugènes exposures.

SUMMARY:
The PIG-A gene (in humans)/Pig-a (in rodents) may be a useful reporter of acquired gene mutation. A simple and reproductive test based on flow cytometry allows detection of Pig-a mutants in a few minutes with low blood volumes. Many studies in rodents showed that detecting Pig-a mutations is useful for identifying genotoxic exposure, but studies are needed in humans to validate this biological marker. The investigators propose to carry out a study to assess the prevalence of PIG-A mutated reticulocytes among 30 patients exposed to genotoxic chemotherapy for breast cancer treatment. The investigators will prospectively collect, for each patient, 4 blood samples of 10mL during chemotherapy: the first one (T0) before chemotherapy (before genotoxic exposure), T1 during treatment (after the third cure), T2 (just at the end of chemotherapy) and T3 (five weeks after the end of chemotherapy). PIG-A mutated cells frequency distributions will be compared between T0, T1, T2 and T3. At the same time, the investigators will document the impact of such a genotoxic exposure using the micronuclei test on in vitro binucleate lymphocytes. The micronuclei test reveals structural or numerical chromosome aberrations caused by aneugenic or clastogenic exposure. This test will be done on T0 and T3 blood samples of each patient.

ELIGIBILITY:
Inclusion Criteria:

* Major patients
* Patients with breast cancer
* Who have benefited from breast surgical treatment and have a poly-chemotherapy adjuvanted by FEC100 and Docetaxel.
* Patients should be able to read and understand French.

Exclusion Criteria:

* Minor Patients
* Pregnant women
* Patients who do not speak French and/or are unable to read and understand French.
* Patients who have had a history of radiotherapy, including those who have received a per-operative radiation therapy as part of the initial management of breast cancer
* Patients who have had a history of chemotherapy outside of the chemotherapy possibly received in the treatment of current breast cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-10 (Actual); Primary Completion 2021-01-10 (Estimated); Study Completion 2021-01-10 (Estimated)

PRIMARY OUTCOMES:
analysis of the frequency of reticulocytes PIG-A mutated | 24 months
  The analyzes will be applied at T0 to determine the intra-assay reproducibility. The frequency distributions of mutated cells will be compared:
  * Between the two groups of patients at T0 then,
  * Within each group between T0 (before exposure), T1 (in process), T2 (end of treatment) and T3 (in therapeutic monitoring post) using non-parametric tests on paired and unpaired.
analysis of the binucleated cell micronuclei frequency in culture | 24 months
  Determining the frequency of micronucleated binucleate cells in culture will be performed on the samples at T0 and T3 each patient of both groups. The frequency distribution of micronucleated cells will be compared within each group between T0 and T3 using non-parametric tests on paired series. A difference shall be considered significant if p <0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Olivier Arnaud, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- : Service de Gynécologie Obstétrique Hôpital Nord, Marseille, Marseille Cedex 20, France